CLINICAL TRIAL: NCT04056780
Title: Diagnosis of Periprosthetic Joint Infection With Synovial Fluid Biomarkers Through Integrated Microfluidic Systems
Brief Title: Integrated Microfluidic Systems for Diagnosis of Periprosthetic Joint Infection
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Chang Gung Memorial Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 201802127B0
Record Dates: First submitted 2019-08-11; First posted 2019-08-14 (Actual); Last update posted 2021-08-03 (Actual); Status verified 2021-07

CONDITIONS: Prosthetic Joint Infection

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Septic group: The septic group will be considered as patients that fulfill the 2018 ICM definition of PJI.
  Interventions: Other: Sample collection study
- Aseptic group: The aseptic group will be considered as patients that don't fulfill the 2018 ICM definition of PJI.
  Interventions: Other: Sample collection study

INTERVENTIONS:
Other: Sample collection study — Sample collection and collection of laboratory values

SUMMARY:
Diagnosing periprosthetic joint infection (PJI) remains a major clinical challenge. The diagnosis of PJI is based on a composition of clinical judgment, serologic test from peripheral blood, synovial fluid cytology and biomarkers, radiography, microbiology, histopathologic evaluation of periprosthetic tissue, and intraoperative findings. The importance of PJI diagnosis give the subsequent treatment options, like the removal of prosthesis, debridement and prosthesis retention and the time of reimplantation.

Currently, The Second International Consensus Meeting (ICM) has announced its criteria for the diagnosis of PJI. The preoperative diagnosis includes serologic tests (C-reactive protein, D-dimer, and erythrocyte sedimentation rate) and synovial fluid biomarkers (white blood cell and differential, leukocyte esterase and ⍺-defensin). The intraoperative diagnosis includes a single positive culture, positive histology, and positive intraoperative purulence. However, some of the markers used in the 2018 ICM criteria, such as ⍺-defensin, leukocyte esterase, and synovial fluid C-reactive protein, are not available in every hospital and cannot be immediately available to clinicians in decision making.

The microfluidic technologies have made a notable impact on the evolution of diagnostic tools by providing a rapid and cost-effective platform for the application of immunoassay techniques. The microfluidic system integrates the complex processing steps of the laboratory protocols into a single chip through logical integration and optimization of processes. Chang Gung Memorial Hospital and National Tsing Hua University have conducted preliminary research to confirm the feasibility of their microfluidic systems.

Therefore, the project will develop a "microfluidic biomarker detection chip" to detect the concentrations three important biomarkers for PJI, including ⍺-defensin, leukocyte esterase and C-reactive protein in synovial fluids. This will be a three-year project. In the 1st year, 50 patients who will be scheduled to undergo unilateral revision total joint arthroplasty (RTJA) will be collected with the synovial fluid and tested on a laboratory platform. In the 2nd year, based on laboratory results, 50 patients undergoing RTJAs will be recruited to develop a microfluidic chip system, and their on-chip performance will be fine-tuned and optimized. In the 3rd year, 50 patients undergoing RTJA will be collected, and the verification of the microfluidic system will be realized. This system will be validated in PJIs cohorts in the first stage of debridement and implant removal, in the interim period, and the second stage of reimplantation. It is expected that biomarker detection chip will improve medical distress and bring important information to clinical decision-making.

ELIGIBILITY:
Inclusion Criteria:

1. Revision total knee arthroplasty
2. Revision total hip arthroplasty
3. Sufficiently annotated clinical and laboratory data for classification by the 2018 ICM criteria for PJI
4. Sufficient synovial fluid for study methods.

Exclusion Criteria:

1. Inadequate synovial fluid for analysis
2. Adverse local tissue reaction (ALTR)
3. Crystalline deposition arthropathy
4. Inflammatory arthropathy flare

Ages: 20 Years to 90 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Given the lack of published data regarding the application of 2nd ICM criteria, we will not perform a power analysis for sample size calculation before the study. All consecutive patients undergoing revision total joint arthroplasty (hips and knees) will be eligible for recruitment.
Sampling Method: Non-Probability Sample
Enrollment: 150 (Estimated)
Dates: Start 2020-04-01 (Actual); Primary Completion 2022-03-31 (Estimated); Study Completion 2022-05-31 (Estimated)

PRIMARY OUTCOMES:
The value of synovial fluid human ⍺-defensin 1-3 (HNP1-3) | Post-operative period after collect per 40 cases (usually within 180-365 days following surgery)
  To test synovial fluid ⍺-defensin
The value of leukocyte esterase (LE) | Immediate post-operative period (usually within 1-2 days following surgery)
  To test synovial fluid LE
The value of synovial C-reactive protein (CRP) | Immediate post-operative period (usually within 1-2 days following surgery)
  To test synovial fluid CRP

CONTACTS AND LOCATIONS:
Locations (1):
- Kaohsiung Chang Gung Memorial Hospital, Kaohsiung City, Taiwan

IPD SHARING:
Plan to Share IPD: No